CLINICAL TRIAL: NCT01947439
Title: Prospective,Multicenter Study of Randomized Comparison of the Biolimus A9-eluting Stent With the Zotarolimus-eluting Stent in Multi-vessel PCI
Brief Title: Comparison of the Biolimus A9-eluting Stent With the Zotarolimus -Eluting Stent in Multi-vessel PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, NAM, Chang-Wook, Associate Professor of Internal Medicine, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BATTLE IN MULTI
Record Dates: First submitted 2013-09-12; First posted 2013-09-20 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Multivessel Coronary Artery Disease
Keywords: multivessel stenting
MeSH Terms: interventions — Percutaneous Coronary Intervention; Biomatrix preparation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biolimus A9 eluting stent (Experimental): biolimus A9 stent( Biomatrix or Biomatrix Flex) will be placed in under Percutaneous Coronary Intervention.
  Interventions: Procedure: Percutaneous Coronary Intervention
- Zotarolimus-eluting stent (Active Comparator): zotarolimus eluting stent (Resolute Integrity) will be placed in under Percutaneous Coronary Intervention.
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Percutaneous Transluminal coronary angioplasty and Intervention will be performed in both of randomized groups of biolimus A9 eluting stent and zotarolimus eluting stent
  Other Names: -Resolute Integrity; -Biomatrix; -Biomatrix Flex

SUMMARY:
The risk of restenosis in the treatment of coronary artery disease has significantly lessened thanks to the introduction of Drug eluting stent.

Yet, debates on the efficacy and safety of stents in complex lesions or patients have been circulated.

Recently, PCI in multiple lesions is universally performed with the development of effective stents in various kinds in the clinics.

However, a randomized study is rare for multi-vessel coronary artery disease in real procedural environments.

The primary purpose of this study is to evaluate the clinical progress of biolimus A9-eluting stent and zotarolimus-eluting stent in multi-vessel coronary artery disease.

DETAILED DESCRIPTION:
The patients who need multi-vessel stenting with multi-vessel coronary artery disease will be enrolled.Each randomization of the enrolled subjects will be done 1:1 (biolimus A9-eluting stent : zotarolimus-eluting stent). Randomization will be stratified by two factors: Diabetes mellitus and Acute coronary syndrome.Clinical follow-up will occur at the following time points; 1 month, 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* patients who need multi-vessel stenting with multi-vessel disease
* patients with signed informed consent

Exclusion Criteria:

* known contraindication to any of the following medications: Aspirin,clopidogrel, heparin, contrast agent, Biolimus or Zotarolimus group
* Cardiogenic shock
* Pregnant women or women with potential childbearing
* End-stage diseases with life expectancy shorter than 2 years
* patients with other Drug eluting stents implanted
* Patients requiring modification of antiplatelet agents for planned major surgery within the first 12 months after the enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 932 (Actual)
Dates: Start 2013-03; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
2-year composite end points | up to 2 years
  All cause death, non fatal myocardial infarction, any revascularization

SECONDARY OUTCOMES:
All cause death | up to 2 years
  All cause death
non-cardiac death | up to 2 years
  non-cardiac death
cardiac death | up to 2 years
  cardiac death
non fatal myocardial infarction | up to 2 years
  non fatal myocardial infarction
Any revascularization | up to 2 years
  Any revascularization
Target lesion revascularization | up to 2 years
  Target lesion revascularization
Target vessel revascularization | up to 2 years
  Target vessel revascularization
stent thrombosis | up to 2 years
  stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Wook Nam, Postdoctoral, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (9):
- South Korea (9):
  - Chonnam National University Hospital, Kwangju, Chonnam
  - Ulsan University Hospital, Ulsan, Gyeongsangbuk-do
  - Inje University Ilsan Paik Hospital, Ilsan, Kyeongki
  - Kosin University Hospital, Busan
  - Daegu Catholic University Medical Center, Daegu
  - Daegu Fatima Hospital, Daegu
  - KyungPook National University Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Lee CH, Lee HJ, Chung TW, Lee S, Hwang J, Kim IC, Cho YK, Yoon HJ, Hur SH, Kim JY, Kim YS, Jang WS, Lee JH, Kim W, Lee JB, Hong YJ, Heo JH, Lee BR, Doh JH, Shin ES, Koo BK, Nam CW. Comparison of Thick Biolimus A9-Eluting Stent and Thin Zotarolimus-Eluting Stent in Multi-Vessel Percutaneous Coronary Intervention. Korean Circ J. 2025 May;55(5):396-407. doi: 10.4070/kcj.2024.0101. Epub 2025 Feb 17. PMID 40097279